CLINICAL TRIAL: NCT04157205
Title: Prospective Evaluation Of Exercise-Induced Cardiac Conduction Instability In Predicting Ventricular Fibrillation Events In Hypertrophic Cardiomyopathy
Acronym: PREDICTVFII
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Imperial College Healthcare NHS Trust (Other); Medtronic (Industry); Barts & The London NHS Trust (Other); Daniel Bagshaw Trust (Unknown); Guy's and St Thomas' NHS Foundation Trust (Other); Brighton and Sussex University Hospitals NHS Trust (Other); University Hospital of Wales (Other); Clinical Research and Trials Unit (Norfolk & Norwich University Hospital, UK) (Other); The Leeds Teaching Hospitals NHS Trust (Other); Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17SM4246
Record Dates: First submitted 2019-11-06; First posted 2019-11-08 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: sudden cardiac arrest; defibrillator
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Death, Sudden, Cardiac

STUDY DESIGN:
Intervention Model Description: Prospective cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Test arm (Experimental): All patients. Single arm study
  Interventions: Diagnostic Test: Non-invasive ECG imaging - CardioInsight test

INTERVENTIONS:
Diagnostic Test: Non-invasive ECG imaging - CardioInsight test — 1. Consent session
  2. Fitting of ECGi vest and CT scan of the chest
  3. Supervised exercise test and Valsalva maneuvre
  4. Programmed stimulation via ICD (selected participants)
  5. Blood tests - genetics

SUMMARY:
Hypertrophic Cardiomyopathy (HCM) is an inherited heart condition. Most people who have it are unaware of any problems relating to it. Unfortunately, a small number of people with the condition can suddenly develop a dangerous fast heart beat that can lead to death. There is no cure, but implanting a cardioverter-defibrillator (ICD), which is like a pacemaker can save the life of affected individuals. However, ICD implantation has its own problems, so choosing who gets an ICD is a very important decision.

The current approach for recommending people for an ICD has limitations and a better method is needed. Investigators have developed a new technique called the 'Ventricular Conduction Stability' (V-CoS). This involves wearing a special vest which records electrical signals from the heart, and then running on a treadmill. Investigators have used it to identify abnormalities in the hearts of people with HCM who have also survived a life-threatening event.

This project aims to test new tool against current methods to ascertain which is better at identifying patients who should have an ICD.

DETAILED DESCRIPTION:
To find out how accurate V-CoS test and other ECGI metrics are, the investigator will study patients with confirmed Hypertrophic Cardiomyopathy currently thought to be high risk. They will be tested by V-CoS and have their conventional risk score worked out. Patients will be followed up currently to 5 years to check if they have had a dangerously fast heartbeat or problems with their defibrillator.

Patients will be recruited primarily from three specialist Inherited Cardiac Diseases clinics in London, but will include other centres as well.

Participants will be interviewed in clinic by our team to explain the study, answer questions and to get permission for the test. Participants can leave the study at any time - it will not affect the way the investigator treat them as patients.

Participants will spend a half day at the Cardiac Investigations unit. This day will consist of, in this order:

1. Any remaining discussion of the study, the tests and the consent needed with the participant.
2. Putting the sensor vest on which will be done by one of the research staff. It looks like a waistcoat with electrical connections and is secured to the patient's skin with conductive jelly underneath to help the recordings.
3. A 3D 'CT' scan of the chest is done to show how the sensor vest lines up with the heart. The scan has a low radiation dose, equivalent to 6 months of natural background radiation.
4. Then the participant will run on the treadmill whilst the vest is used to take recordings. The lowest V-CoS test score will be recorded from each participant and used to predict their risk.
5. Participants will have the V-CoS test repeated whilst doing the Valsalva maneuver. This is when participant attempt to blow out as much air as possible from lungs, but without letting any out from mouth or nose.
6. Participants with implanted pacemakers or defibrillators may undergo a test where the investigator give them extra heartbeats using their implanted device. The sensor vest will be used to take recordings. The investigator want to see if V-CoS scores can be lowered further than with exercise testing.
7. Participants will have a blood test or cheek swab to send for genetic testing. Then participants will be followed up. If they have a defibrillator they will be telephoned and seen in the ICD clinic every 6 months. If they do not have a defibrillator they will get follow up by telephone every 3 months. Maximum follow up is 5 years.

The results will be looked at by independent researchers to reduce bias.

ELIGIBILITY:
Inclusion criteria

* Does the patient have maximum wall thickness >13mm by any imaging technique? i) If so, does the patient have a first degree relative (sibling, parent, child) with a formal diagnosis of HCM -AND- ii) Does the patient have any of the following: Does the patient have any of the following: abnormal Doppler myocardial imaging or strain, incomplete systolic anterior motion, elongation of mitral valve leaflets and abnormal papillary muscles, abnormal ECG? -OR-
* Does the patient have maximum wall thickness 15mm or more by any imaging technique?
* Is the patient male or female 18-100years of age?
* High or intermediate risk for sudden cardiac death from HCM based on the ESC risk calculator predicting >4% risk over 5 years by specialist inherited cardiac disease clinic. This would use the online SCD-risk calculator

Exclusion criteria

* Patients with previous cardiac arrest
* Patients with haemodynamically unstable VT needing medical attention.
* Evidence of one of the following conditions causing secondary hypertrophy:

  a. Hypertension >200/100; Severe aortic stenosis; Anderson-Fabry disease; Myocarditis; Congenital heart disease; TTR-related amyloidosis; Myotonic dystrophy; Mitochondrial disease, Noonan syndrome, LEOPARD syndrome, Costello syndrome, Danon disease, Friedreich's ataxia, Glycogen storage disease, FHLI mutation, PRKAG2 mutations
* Patients with previous appropriate therapy from an ICD.
* Patients under the age of 18 years
* Patients who are not safe to discontinue Beta blockers
* Patients unable to exercise due to musculoskeletal problems
* Patients with skin allergies to ECG gel/electrodes.
* Life expectancy shorter than the duration of the trial.
* Pregnant or planning pregnancy at the time of CT scan.
* Patients unable to consent to the study protocol or provide contact details for follow up.
* Patients currently participating in an interventional medical or device trial.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2019-11-10 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with sudden cardiac death, or appropriate therapy from ICD for VT/VF. | 5 years
  Sudden cardiac death, or appropriate therapy from ICD for VT/VF follow up assessed by phone call to study participant

SECONDARY OUTCOMES:
Number of Participants with syncopal events of unknown cause in patients without ICDs | 5 years
  syncopal events of unknown cause in patients without ICDs
Number of Participants with inappropriate therapy from ICD | 5 years
  inappropriate therapy from ICD
Number of Participants with indeterminate therapy from ICD | 5 years
  indeterminate therapy from ICD
Number of Participants with complications from ICD implant | 5 years
  complications from ICD implant
Number of Participants with complications from performing V-CoS test | 5 years
  complications from performing V-CoS test

CONTACTS AND LOCATIONS:
Overall Officials: Prapa Kanagaratnam, FRCP, PhD, Principal Investigator — Imperial College NHS Trust
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Participating sites will have access to the all the anonymised clinical data after completion for subtudies.